CLINICAL TRIAL: NCT06173973
Title: Effects of Ketone Supplementation on Acute Alcohol Withdrawal Symptoms During Alcohol Withdrawal Management
Brief Title: Effects of Ketone Supplementation on Acute Alcohol Withdrawal
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Corinde Wiers, PhD, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 854682
Record Dates: First submitted 2023-11-28; First posted 2023-12-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal; Alcohol Dependence; Ketosis
Keywords: Alcohol Use Disorder; Alcohol Withdrawal; Alcohol Dependence; Ketone Supplement; Ketosis
MeSH Terms: conditions — Alcoholism; Ketosis

STUDY DESIGN:
Intervention Model Description: Placebo controlled, Double blinded study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketone Supplement (Active Comparator): Ketone Supplement drink with 10 g ketones three times daily for five days.
  Interventions: Dietary Supplement: Kenetik; Ketone Concentrate
- Placebo Beverage (Placebo Comparator): Matching Placebo drink three times daily for five days
  Interventions: Dietary Supplement: Isocaloric dextrose placebo

INTERVENTIONS:
Dietary Supplement: Kenetik; Ketone Concentrate — Ketone Supplement
  Other Names: D-hydroxybutyric acid and R-1,3 butanediol
  Arms: Ketone Supplement
Dietary Supplement: Isocaloric dextrose placebo — Drink that is taste and visually matched to Ketone supplement
  Arms: Placebo Beverage

SUMMARY:
The goal of this study is to study the effects of the ketone supplement Kenetik compared to placebo (an inactive beverage) on alcohol withdrawal symptoms during the 5 days of clinical alcohol withdrawal management treatment at the Caron Treatment Center.

DETAILED DESCRIPTION:
This is a 5 day double-blinded, placebo-controlled intervention study of 50 treatment-seeking individuals with AUD, who are receiving detoxification treatment at Caron Treatment Center. Participants will be recruited for participation within 48 hours of admission to the inpatient unit. Participants will be consented and randomized to receive 10 g of ketone supplement three times daily (n=30; 1,3-butanediol and D-hydroxybutyric acid from Kenetik, VitaNav Inc., Washington D.C.) for 5 days or a placebo beverage (n=20). Benzodiazepines and other "comfort" medications will be administered daily following the Caron withdrawal management protocol, with additional benzodiazepines administered based on withdrawal symptoms, monitored with the revised Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar). The CIWA-Ar is given three or more times per day clinically to determine patient withdrawal levels and adjust medication dosages. Total daily maximum CIWA-Ar scores, benzodiazepine dosage and other "comfort" medications will be analyzed with a repeated measures design, with a binary factor for intervention, factor of time, and intervention by time interaction. Daily mood and alcohol craving questions will assess differences between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

1. Meets current DSM-5 criteria for AUD and admitted for alcohol withdrawal management treatment at Caron Treatment Center
2. Willingness to provide signed, informed consent and commit to completing the procedures in the study

Exclusion Criteria:

1. Current, gastrointestinal (GI), liver or other clinically significant physical disease that may interfere with the intake of the Ketone Supplement based on medical history, and evaluation of the Study Physician.
2. Currently pregnant or lactating, based on urine pregnancy test and clinical exam.
3. Current significant withdrawal from other substances, including benzodiazepines, opioids that require medication management for withdrawal and may interfere with study results/withdrawal management plan.
4. Judged by the principal investigator, Study Physician, or their designee to be an unsuitable candidate for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Effects of ketone supplement Kenetik, three times daily (TID), versus placebo, on the need for benzodiazepines (daily use in mg). | 5 days
  To examine the effects of ketone supplement Kenetik, three times daily (TID), versus placebo, on the need for benzodiazepines (daily use in mg), while undergoing inpatient acute withdrawal management.

SECONDARY OUTCOMES:
Effects of ketone supplement Kenetik, three times daily (TID), versus placebo, on Clinical Institute Withdrawal Assessment Alcohol Scale Revised (CIWA-Ar) scores (daily maximum scores). | 5 days
  To examine the effects of ketone supplement Kenetik, three times daily (TID), versus placebo, on Clinical Institute Withdrawal Assessment Alcohol Scale Revised (CIWA-Ar) scores (daily maximum scores, range 0-67) while undergoing inpatient acute withdrawal management.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde E Wiers, Ph.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Pennsylvania Center for Studies of Addiction, Philadelphia, Pennsylvania
  - Caron Treatment Center, Wernersville, Pennsylvania